CLINICAL TRIAL: NCT06640127
Title: A Randomized Comparative Study on Internal Sinus Lifting With Simultaneous Implant Placement Using Two Different Techniques
Brief Title: Use of Specifically Designed Drills for Internal Sinus Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Associated Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-4.1/30; 23834 (Other Grant/Funding Number: Ege University)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vertical Alveolar Bone Loss; Sinus Lifting; Implant Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Sinus lifting and implant placement with osteotomes
  Interventions: Procedure: Sinus lifting and implant placement with osteotomes
- Test Group (Experimental): Sinus lifting and implant placement with specifically designed drills
  Interventions: Procedure: Sinus lifting and implant placement with specifically designed drills

INTERVENTIONS:
Procedure: Sinus lifting and implant placement with osteotomes — Osteotomes with increasing diameters were used for sinus membrane elevation and implant insertion
  Arms: Control Group
Procedure: Sinus lifting and implant placement with specifically designed drills — Sequential drills were used for sinus membrane elevation and implant insertion
  Arms: Test Group

SUMMARY:
This study was conducted at Ege University, School of Dentistry, Izmir, Turkey. Patients enrolled require implant placement to the atrophic posterior maxilla. Patients were treated with either the specifically designed drills or the osteotomes. The outcome variables were primary stability, marginal bone loss, implant survival, and patient-reported outcomes. The investigators aimed to compare the treatment outcomes of two different techniques used in dental implant placement with internal sinus lifting.

DETAILED DESCRIPTION:
This prospective, randomized clinical study was conducted at the Ege University School of Dentistry and Department of Oral and Maxillofacial Surgery. Patients with atrophic maxillas and at least one tooth loss in this region were included. Randomization was performed to assign the patients to study groups. Patients treated with internal sinus lift using osteotome and implant surgery were assigned to Group 1, and patients treated with internal sinus lift using specifically designed drills and implant surgery were assigned to Group 2. At six months postoperatively, the healing cap was inserted during the second stage of surgery.

All implants were assessed based on primary stability (using implant stability quotient and torque value), marginal bone loss (as millimeters), and implant survival (as a percentage). Also, patient-reported outcomes were collected, including pain (using a visual analog scale), analgesic consumption (number of drugs taken during a week), and oral health impact profile survey).

ELIGIBILITY:
Inclusion Criteria:

* Unilaterally or bilaterally missing teeth in the posterior maxilla,
* Residual bone height (4 mm to 6 mm),
* Completed periodontal and oral hygiene treatment,
* American Society of Anesthesiologists (ASA) score of I or II,
* > 18 years old,
* Willingness to participate

Exclusion Criteria:

* Infection or pathology related to maxillary sinus and surgical site,
* Tooth extraction within six months in the surgical site,
* Previous maxillary sinus surgery,
* Parafunction,
* Medical conditions associated with impaired or delayed wound healing,
* Smoking habit and alcohol or drug abuse,
* Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Mean of implant insertion quantity (ISQ) value | at surgery
  Calculation of ISQ value for each implant
Mean of torque value | at surgery
  Calculation of torque value for each implant

SECONDARY OUTCOMES:
Marginal bone loss | through study completion, an average of 1 year
  Change in peri-implant bone level
Implant survival | through study completion, an average of 1 year
  Number of mobil or loss implants
Pain Score | at postoperative first week
  Pain level recorded between 0 to 10 points
Analgesic consumption | at postoperative first week
  Number of analgesic taken on a daily basis
Oral health impact profile questionnaire | preoperatively, at postoperative first week, and at postoperative 6 months
  Total score of self-administered questionnaire assessed using Likert-point scale between 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Işık, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No